CLINICAL TRIAL: NCT04557982
Title: Creating a Czech Version of the Simplified Faces Pain Scale and the Simplified Concrete Ordinal Pain Scale
Status: Completed | Type: Observational
Sponsor: Palacky University (Other)
Collaborators: University of Pardubice (Other)
Responsible Party: Principal Investigator, Petra Kasparova, Principal Investigator, Palacky University
Other Study IDs: 123
Record Dates: First submitted 2020-08-28; First posted 2020-09-22 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Pain Measurement
Keywords: Pain Measurement; Pain Assessment; Nurse; Nursing; Child; Pediatrics; Instrument; Scale; Tool

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Children aged 3 < 4 years: Children aged 3 < 4 years will be recruited using convenience sampling and meeting the inclusion criteria (child Czech-speaking, able to distinguish between small/medium sized/large toy, willing to cooperate, parent/significant other is present and signs informed consent). The child will be explained the use of the S-COS, and S-FPS and self-reports pain intensity immediately prior to the procedure (Time 0), immediately after the procedure (Time 1) and after 5-10 minutes (Time 2). Furthermore, at Time 0, 1 and 2, the child´s pain level is independently assessed by the attending nurse and by the researcher.
  Interventions: Procedure: A painful procedure (peripheral venepuncture)
- Children aged 4 < 5 years: Children aged 4 < 5 years will be recruited using convenience sampling and meeting the inclusion criteria (child Czech-speaking, able to distinguish between small/medium sized/large toy, willing to cooperate, parent/significant other is present and signs informed consent). The child will be explained the use of the S-COS, and S-FPS and self-reports pain intensity immediately prior to the procedure (Time 0), immediately after the procedure (Time 1) and after 5-10 minutes (Time 2). Furthermore, at Time 0, 1 and 2, the child´s pain level is independently assessed by the attending nurse and by the researcher.
  Interventions: Procedure: A painful procedure (peripheral venepuncture)
- Children aged 5 < 6 years: Children aged 5 < 6 years will be recruited using convenience sampling and meeting the inclusion criteria (child Czech-speaking, able to distinguish between small/medium sized/large toy, willing to cooperate, parent/significant other is present and signs informed consent). The child will be explained the use of the S-COS, and S-FPS and self-reports pain intensity immediately prior to the procedure (Time 0), immediately after the procedure (Time 1) and after 5-10 minutes (Time 2). Furthermore, at Time 0, 1 and 2, the child´s pain level is independently assessed by the attending nurse and by the researcher.
  Interventions: Procedure: A painful procedure (peripheral venepuncture)

INTERVENTIONS:
Procedure: A painful procedure (peripheral venepuncture) — The child will undergo a peripheral venepuncture during a scheduled visit to a hospital clinic and routinely provided care.

SUMMARY:
The aim is to create a Czech version of pain assessment tools in children, the Simplified Faces Pain Scale (S-FPS) and the Simplified Concrete Ordinal Scale (S-COS), including methodology for their use in practice, and to establish their validity and reliability in pre-school children. The S-FPS is composed of three faces representing three different levels of pain, and the S-COS shows three blocks that symbolize three levels of intensity of pain. The instrument translation and linguistic validation process will be based on the International Society for Pharmacoeconomics and Outcomes Research guidelines (Wild et al., 2005). Validity and reliability will be tested by comparing the children´s pain intensity using the S-FPS and S-COS, which will be completed by the children, and the instrument Face, Legs, Activity, Cry, Consolability (FLACC), which will be completed independently by the attending nurse and the researcher. A repeated measures design will be used as all assessments will be performed prior to a painful procedure (peripheral venepuncture) and will be repeated twice after the painful procedure, once immediately after the painful procedure and a second time 5-10 minutes after the painful procedure. A total of 180 children with will be recruited (aged 3-6 years) from whom complete data will be obtained.

DETAILED DESCRIPTION:
Introduction:

For a long time, there has been a myth that children do not remember pain that they were subjected to in the past. However, it has been confirmed that children transfer their negative experience of pain to adulthood. As many studies have shown, information about pain can be obtained from patient self-report, physical response and/or behavioral manifestations. Self-report is considered as the gold standard. The major problem is that most preschool-aged children do not have the necessary cognitive development to use the standard scales.

A group of experts in Canada has developed two new pain scales for this particular age, the Simplified Faces Pain Scale (S-FPS) and the Simplified Concrete Ordinal Scale (S-COS). The S-FPS consists of three faces representing three levels of pain intensity, and the S-COS consists of three blocks that symbolize pain intensity, ranging from mild pain (one block) to severe pain (three blocks). Their research was based on the assumption that younger children are able to distinguish only two or three levels of pain intensity.

Aim:

The aim is to create a Czech version of pain assessment tools in children, the Simplified Faces Pain Scale (S-FPS) and the Simplified Concrete Ordinal Scale (S-COS), including methodology for their use in practice, and to establish their validity and reliability in pre-school children.

The cognitive ability of the child for the research study will be verified by two control tasks, presented to each child prior to enrolment:

"Describe the presented toy (a star). Choose the biggest star from these three toys (stars) of different sizes."

The tools and procedure:

Children will be asked to evaluate their pain intensity using the S-FPS and the S-COS on three different occasions linked to a painful procedure (before peripheral venepuncture, immediately after the peripheral venepuncture and 5-10 minutes after the peripheral venepuncture).

Before the first venepuncture, the researcher will ask the parents what specific word their child uses to describe pain and then asks the child: "Do you have any pain?," (the child´s word used for pain). If the answer is "no", then the researcher writes "0". If he/she responds "yes", then the child is asked to allocate the perceived pain intensity to the picture, i.e. a corresponding face using the S-FPS, and a corresponding number of blocks, using the S-COS.

The researcher and the attending nurse evaluate the pain at each of these time points using the behavioral scale Face, Legs, Activity, Cry, Consolability (FLACC) (Merkel et al., 2002). The child, the researcher and the attending nurse will do their assessment independently.

Characteristics of the respondents:

The research group will consist of a total of 180 pre-school children (with complete data on all items) who will be subjected to a peripheral venepuncture during their visit to a hospital clinic and who have not received any analgesia prior to the procedure (the researcher will obtain this information during the interview with the parents).

Data Collection:

Before collecting the data, the researcher will individually explain the whole procedure to all participants in such a way that they understand it well, especially to children with regard to their cognitive development. Furthermore, the attending nurse will undergo training concerning data collection and the entire study, as well.

The researcher personally contacts the parents of the child and the child in the waiting room of the Children's Clinic in a tertiary hospital in the city of Olomouc and informs them of the research project. If they agree to being enrolled, the child will be screened for sufficient cognitive development and ability to distinguish three different sizes. This will be done using three identical toys (different sizes) that will be presented to the child and the researcher asks him/her to order the toys from the smallest to the largest. The correct arrangement of toys is the basic criterion for inclusion in the study. The child, the researcher and the attending nurse (the research assistant) participate in the pain assessment. Parents will stay with the child during the whole process, but they do not evaluate the pain. They will be instructed not to provide the child with any verbal or behavioural cues or engage in any behaviour that would either distract the child or that would affect the child´s performance during data collection.

The research study is divided into 3 phases:

Phase 1: before peripheral venepuncture: The researcher and the attending nurse complete an observational pain report using the FLACC. The child assesses if he/she has pain. If the answer is "no", the researcher writes "0", if the response is "yes", the child will evaluate pain using each self-report tool (S-FPS and S-COS).

Phase 2: immediately after peripheral venepuncture: The researcher and nurse complete an observational pain report using the FLACC. The child assesses if he/she has pain. If the answer is "no", the researcher writes "0", if the response is "yes", the child will evaluate pain using each self-report tool (S-FPS and S-COS).

Between phase 2 and phase 3, the child is distracted from the procedure. He/she may play with the parent etc.

Phase 3: 5-10 min. after peripheral venepuncture: The researcher and nurse complete an observational pain report using the FLACC. The child assesses if he/she has pain. If the answer is "no", the researcher writes "0", if the response is "yes", the child will evaluate pain using each self-report tool (S-FPS and S-COS).

Randomization:

Each child evaluates pain using both the S-FPS and S-COS. The order in which these two tools are presented to the child will be random. Randomization will be done for each child three times, before phase 1, phase 2 and phase 3. The order is randomly assigned by a computer program (www.randomizer.org).

ELIGIBILITY:
Inclusion Criteria:

* Czech-speaking
* male or female
* aged 3-6 years
* scheduled to undergo peripheral venepuncture
* ability to distinguish three sizes using a toy: small/medium sized/large
* signed informed consent by parent/significant other

Exclusion Criteria:

* non-Czech speaking
* refusal to cooperate by the child,
* low cognitive ability (inability to distinguish three sizes using a toy: small/medium sized/large)
* refusal to cooperate by the parent/significant other

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Subjects indicated for peripheral venepuncture (blood draw or peripheral IV cannulation)
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Pain intensity at Time 0 (immediately prior to the painful procedure) using the Simplified Faces Pain Scale (using self-report). | Time 0 (immediately prior to the painful procedure)
  The Simplified Faces Pain Scale is a self-report measure of pain intensity consisting of pictures of three faces printed on a form, each face represents a different level of pain. Beginning from the left, the first face = mild pain, the middle face = moderate pain, the last face = severe pain.
Pain intensity at Time 0 (immediately prior to the painful procedure) using the Simplified Concrete Ordinal Scale (using self-report). | Time 0 (immediately prior to the painful procedure)
  The Simplified Concrete Ordinal Scale is a self-report measure of pain intensity consisting of three blocks that symbolize pain intensity, ranging from mild pain (one block) to severe pain (three blocks).
Pain intensity at Time 0 (immediately prior to the painful procedure) using the The Face, Legs, Activity, Cry, Consolability instrument (using proxy report by the researcher). | Time 0 (immediately prior to the painful procedure)
  The Face, Legs, Activity, Cry, Consolability scale is an observational (behavioral) instrument used to assess pain using 5 criteria: the face, legs, activity, cry, and consolability, which are each assigned a score of 0, 1, or 2. Total score ranges from 0-10 with 10 representing the most severe pain possible.
Pain intensity at Time 0 (immediately prior to the painful procedure) using the The Face, Legs, Activity, Cry, Consolability instrument (using proxy report by the attending nurse). | Time 0 (immediately prior to the painful procedure)
  The Face, Legs, Activity, Cry, Consolability scale is an observational (behavioral) instrument used to assess pain using 5 criteria: the face, legs, activity, cry, and consolability, which are each assigned a score of 0, 1, or 2. Total score ranges from 0-10 with 10 representing the most severe pain possible.
Pain intensity at Time 1 (immediately after the painful procedure) using the Simplified Faces Pain Scale (using self-report). | Time 1 (immediately after the painful procedure)
  The Simplified Faces Pain Scale is a self-report measure of pain intensity consisting of pictures of three faces printed on a form, each face represents a different level of pain. Beginning from the left, the first face = mild pain, the middle face = moderate pain, the last face = severe pain.
Pain intensity at Time 1 (immediately after the painful procedure) using the Simplified Concrete Ordinal Scale (using self-report). | Time 1 (immediately after the painful procedure)
  The Simplified Concrete Ordinal Scale is a self-report measure of pain intensity consisting of three blocks that symbolize pain intensity, ranging from mild pain (one block) to severe pain (three blocks).
Pain intensity at Time 1 (immediately after to the painful procedure) using the The Face, Legs, Activity, Cry, Consolability instrument (using proxy report by the researcher). | Time 1 (immediately after the painful procedure)
  The Face, Legs, Activity, Cry, Consolability scale is an observational (behavioral) instrument used to assess pain using 5 criteria: the face, legs, activity, cry, and consolability, which are each assigned a score of 0, 1, or 2. Total score ranges from 0-10 with 10 representing the most severe pain possible.
Pain intensity at Time 1 (immediately after to the painful procedure) using the The Face, Legs, Activity, Cry, Consolability instrument (using proxy report by the attending nurse). | Time 1 (immediately after the painful procedure)
  The Face, Legs, Activity, Cry, Consolability scale is an observational (behavioral) instrument used to assess pain using 5 criteria: the face, legs, activity, cry, and consolability, which are each assigned a score of 0, 1, or 2. Total score ranges from 0-10 with 10 representing the most severe pain possible.
Pain intensity at Time 2 (5-10 minutes after the painful procedure) using the Simplified Faces Pain Scale (using self-report). | Time 2 (immediately after the painful procedure)
  The Simplified Faces Pain Scale is a self-report measure of pain intensity consisting of pictures of three faces printed on a form, each face represents a different level of pain. Beginning from the left, the first face = mild pain, the middle face = moderate pain, the last face = severe pain.
Pain intensity at Time 2 (5-10 minutes after the painful procedure) using the Simplified Concrete Ordinal Scale (using self-report). | Time 2 (5-10 minutes after the painful procedure)
  The Simplified Concrete Ordinal Scale is a self-report measure of pain intensity consisting of three blocks that symbolize pain intensity, ranging from mild pain (one block) to severe pain (three blocks).
Pain intensity at Time 2 (5-10 minutes after to the painful procedure) using the The Face, Legs, Activity, Cry, Consolability instrument (using proxy report by the researcher). | Time 2 (5-10 minutes after the painful procedure)
  The Face, Legs, Activity, Cry, Consolability scale is an observational (behavioral) instrument used to assess pain using 5 criteria: the face, legs, activity, cry, and consolability, which are each assigned a score of 0, 1, or 2. Total score ranges from 0-10 with 0 representing no pain.
Pain intensity at Time 2 (5-10 minutes after to the painful procedure) using the The Face, Legs, Activity, Cry, Consolability instrument (using proxy report by the attending nurse). | Time 2 (5-10 minutes after the painful procedure)
  The Face, Legs, Activity, Cry, Consolability scale is an observational (behavioral) instrument used to assess pain using 5 criteria: the face, legs, activity, cry, and consolability, which are each assigned a score of 0, 1, or 2. Total score ranges from 0-10 with 0 representing no pain.

CONTACTS AND LOCATIONS:
Overall Officials: Petra Kašparová, Mgr., Principal Investigator — Palacky University
Locations (1):
- University Hospital Olomouc, Olomouc, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Emmott AS, West N, Zhou G, Dunsmuir D, Montgomery CJ, Lauder GR, von Baeyer CL. Validity of Simplified Versus Standard Self-Report Measures of Pain Intensity in Preschool-Aged Children Undergoing Venipuncture. J Pain. 2017 May;18(5):564-573. doi: 10.1016/j.jpain.2016.12.015. Epub 2017 Jan 6. PMID 28069521
- [Background] Merkel S, Voepel-Lewis T, Malviya S. Pain assessment in infants and young children: the FLACC scale. Am J Nurs. 2002 Oct;102(10):55-8. doi: 10.1097/00000446-200210000-00024. No abstract available. PMID 12394307
- [Background] Wild D, Grove A, Martin M, Eremenco S, McElroy S, Verjee-Lorenz A, Erikson P; ISPOR Task Force for Translation and Cultural Adaptation. Principles of Good Practice for the Translation and Cultural Adaptation Process for Patient-Reported Outcomes (PRO) Measures: report of the ISPOR Task Force for Translation and Cultural Adaptation. Value Health. 2005 Mar-Apr;8(2):94-104. doi: 10.1111/j.1524-4733.2005.04054.x. PMID 15804318
- See also: Research Randomizer — https://www.randomizer.org/